CLINICAL TRIAL: NCT01281774
Title: An Adaptive, Phase I, Randomised, Placebo-controlled, Sponsor-unblinded, Multiple Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of Intravenous CSL112 in Healthy Volunteers
Brief Title: A Multiple Ascending Dose Study of CSL112 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSLCT-HDL-10-68
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
MeSH Terms: interventions — CSL112

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CSL112 (Experimental): Multiple ascending intravenous doses of CSL112
  Interventions: Biological: CSL112
- Placebo (Placebo Comparator): Multiple intravenous infusions of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CSL112 — reconstituted high density lipoprotein
  Arms: CSL112
Biological: Placebo — Normal saline (0.9%)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of CSL112 in healthy volunteers after multiple infusions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 18 years to less than 55 years
* Body weight 50kg or greater
* Body mass index (BMI) between 18 and 42.0 kg/m2

Exclusion Criteria:

* Evidence of a clinically significant medical condition, disorder or disease
* Evidence of hepatobiliary disease
* Any clinically relevant abnormal laboratory test result
* Evidence or history of alcohol or substance abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The frequency of drug-related adverse events | Up to 6 days after each infusion
The frequency of redness and swelling at the infusion site | up to 24 hours after each infusion
Clinically important elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) | up to 6 days after each infusion

SECONDARY OUTCOMES:
Pharmacokinetic profile of apoA-I after multiple intravenous infusions | up to 7 days after each infusion

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Cardiovascular, Study Director — CSL Limited
Locations (1):
- Q-Pharm, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] Zheng B, Duffy D, Tricoci P, Kastrissios H, Pfister M, Wright SD, Gille A, Tortorici MA. Pharmacometric analyses to characterize the effect of CSL112 on apolipoprotein A-I and cholesterol efflux capacity in acute myocardial infarction patients. Br J Clin Pharmacol. 2021 Jun;87(6):2558-2571. doi: 10.1111/bcp.14666. Epub 2020 Dec 23. PMID 33217027
- [Derived] Easton R, Gille A, D'Andrea D, Davis R, Wright SD, Shear C. A multiple ascending dose study of CSL112, an infused formulation of ApoA-I. J Clin Pharmacol. 2014 Mar;54(3):301-10. doi: 10.1002/jcph.194. Epub 2013 Oct 22. PMID 24122814